CLINICAL TRIAL: NCT06976034
Title: oCular Examination at Cell RESolution With Optical TransmissionTomography
Acronym: CERES-OTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P24-01
Record Dates: First submitted 2025-05-02; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma Associated With Other Ocular Disorders
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Prospective, exploratory, longitudinal, non-randomized, single-center study including patients and healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Ocular Disease (Experimental): Patients: an imaging examination by each system (OTT + OCT + specular microscopy) will be carried out by two different operators, and several imaging images will be taken from different positions. These examinations will be performed at the inclusion visit and at follow-up visits as part of the usual management of the disease up to a maximum of 4 years
  Interventions: Device: Optical Transmission Tomography (OTT); Device: Optical Coherence Tomography (OCT); Device: Specular Microscopy (SM)
- Healthy volunteers (Active Comparator): Healthy Volunteers: an imaging examination by each system (OTT + OCT + specular microscopy) will be carried out twice, at the inclusion visit and at 24 months (2 years), the maximum duration of participation for healthy volunteers. Several imaging sessions will be carried out by two different operators at different positions
  Interventions: Device: Optical Transmission Tomography (OTT); Device: Optical Coherence Tomography (OCT); Device: Specular Microscopy (SM)

INTERVENTIONS:
Device: Optical Transmission Tomography (OTT) — Multiple imaging sessions added by research using the systems described (OTT) will be carried out by two different operators at different positions during these sessions.
Device: Optical Coherence Tomography (OCT) — Multiple imaging sessions (OCT) already used in standard of care will be performed by two different operators at different positions during these sessions.
Device: Specular Microscopy (SM) — Multiple imaging sessions (SM) already used in standard of care will be performed by two different operators at different positions during these sessions.

SUMMARY:
Understanding the pathogenesis of eye diseases has benefited greatly from recent advances in ophthalmic imaging. However, current clinical imaging systems, such as optical coherence tomography (OCT), are limited in terms of resolution, acquisition speed or access to certain eye functions. Our team has participated in the development of a new generation of imaging technology known as optical transmission tomography (OTT), which enables imaging of the anterior parts of the eye with high cellular resolution, a wide field of view and reduced examination delay.

DETAILED DESCRIPTION:
For healthy subjects: an imaging examination using each system (OTT + OCT + specular microscopy) will be carried out twice, at an interval of two (2) years (inclusion visit + visit at 24 months). Several imaging images will be taken by two different operators during these sessions.

For patients: an imaging examination using each system (OTT + OCT + specular microscopy) will be carried out by two different operators, and several imaging images will be taken. These examinations will be carried out at the inclusion visit and at the following visits according to the disease assessment schedule, lasting up to a maximum of 4 years.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* 200 subjects aged 18 to 80 years;
* Male or female;
* with an ocular disease affecting the cornea, ocular surface, lens (cataract) or glaucoma, or requiring refractive surgery or post-refractive surgery follow-up;
* Are covered by the French Assurance Maladie;
* Have signed an express, free and informed consent form.

For Healthy volunteers:

* 100 subjects aged 18 to 80 years;
* Male or female;
* Healthy subjects with no known pathology directly or indirectly affecting ocular structures;
* Covered by the French Assurance Maladie.
* Having signed an express, free and informed consent form.

Exclusion Criteria:

For all participants:

* Inability to hold a still position on a standard ophthalmic chin rest;
* Conjunctivitis or other contagious contact disease in active phase;
* Having an implanted pacemaker or other electronic medical device;
* Having a predisposition to iridocorneal angle closure;
* Vulnerable persons or persons under legal protection (pregnant or breast-feeding women; persons under guardianship,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2029-11-12 (Estimated); Study Completion 2029-11-12 (Estimated)

PRIMARY OUTCOMES:
Image quality | between 1 day and 4 years
  Quality assessed by two blinded experts.
  This is an evaluation of image quality in terms of operation according to the following scheme.
  Quality assessment:
  - Sufficient quality : Yes Or No
  If no, tick yes, below and fill in the cause:
  Insufficient quality: ☒ yes ☐ no
  Cause:
  * Technical problem Or
  * Patient-related problem (inability to fix, or comply with procedure, etc.)
Endothelial cell density | between 1 day and 4 years
  Assessment of endothelial cell density.
Imaging new corneal and lens structures | between 1 day and 4 years
  corneal and lens structures:measure density in other cell types

CONTACTS AND LOCATIONS:
Overall Officials: Nacim BOUHERAOUA, PU-PH, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France